CLINICAL TRIAL: NCT02821624
Title: First-in-Human Phase 1 Safety, Pharmacokinetic, and Food Effect Study of Single Ascending Doses of G1T38 in Healthy Male and Female Subjects
Brief Title: First-in-Human Safety, PK, and Food Effect Study of Single Ascending Doses of G1T38 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: G1T38-01; 2016-001201-17 (EudraCT Number)
Record Dates: First submitted 2016-06-28; First posted 2016-07-01 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort 1 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 2 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 3 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 4 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 5 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 6 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 7 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 8 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 9 - Food Effect (Experimental): G1T38
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor)
- Cohort 10 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 11 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo
- Cohort 12 (Experimental): G1T38 or placebo
  Interventions: Drug: G1T38 (CDK 4/6 Inhibitor); Drug: Placebo

INTERVENTIONS:
Drug: G1T38 (CDK 4/6 Inhibitor) — CDK 4/6 Inhibitor
  Other Names: G1T38
Drug: Placebo — Placebo
  Arms: Cohort 1; Cohort 10; Cohort 11; Cohort 12; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7; Cohort 8

SUMMARY:
This first-in-human (FIH) study will provide the first safety and pharmacokinetic (PK) data for G1T38 in humans and will allow further development of G1T38 in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 40-65 years of age; no clinically significant findings reported following detailed physical examination, medical history, vital signs, clinical laboratory tests, and ECGs as deemed by the PI
* Body mass index (BMI) in the range of 18 to 32 kg/m2 (inclusive) at screening, and weighing at least 50 kg
* Nonusers of nicotine-containing products for at least the previous 3 months prior to dosing or nonsmokers
* Agreement to use birth control during the study and 3 months post last visit.
* Able to comply with all protocol requirements and procedures

Exclusion Criteria:

* Clinically significant abnormalities found during physical examinations, medical history review, ECGs (QTcF interval > 450 milliseconds for males and >470 milliseconds for females), vital signs, and laboratory tests (including positive HIV, hepatitis B and C)
* Participated in in a previous clinical study with an investigational product in the last 60 days
* History of any serious allergic reaction to any medication
* Any blood or plasma donation or other loss of blood at a volume exceeding 500 mL within 3 months before dosing
* History of drug or alcohol abuse in the last 2 years
* Pregnant or lactating women
* Any other issues which, in the opinion of the PI, will make the subject ineligible for study participation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12-15 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Related Adverse Event, including Abnormal Laboratory Events | Up to Day 7
  All AEs, including clinical laboratory, vitals signs, physical examinations and ECGs will be analyzed in all subjects receiving study drug through 7 days post dose of study drug.

SECONDARY OUTCOMES:
Pharmacokinetics of G1T38: Maximum Plasma Concentration (Cmax) | Day 1, 2, 3, 4 and 5
  The observed peak plasma concentration determined from the plasma
Pharmacokinetics of G1T38: Area under Curve - plasma concentration (AUC) | Day 1, 2, 3, 4 and 5
  Area under the plasma concentration-time curve
Pharmacokinetics of G1T38: Plasma: terminal half life (T1/2) | Day 1, 2, 3, 4 and 5
  G1T38: Plasma- terminal half life (T1/2)
Pharmacokinetics of G1T38: Plasma - Volume of distribution | Day 1, 2, 3, 4 and 5
  Volume of distribution in the terminal elimination phase

CONTACTS AND LOCATIONS:
Overall Officials: Regner Tiessen, MD, Principal Investigator — PRA Early Development Clinic
Locations (1):
- PRA Early Development Clinic, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided